CLINICAL TRIAL: NCT01571349
Title: Hemostasis in Patients With Idiopathic Thrombocytopenic Purpura
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Gaab Soo Kim, Professor, Samsung Medical Center
Other Study IDs: 2012-02--85-001
Record Dates: First submitted 2012-04-02; First posted 2012-04-05 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: rebalanced hemostasis; idiopathic thrombocytopenic purpura; coagulation status
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- chronic ITP group: ITP patients with elevated level of vWF, ITP patients with preserved MA of thromboelastography
- acute ITP group: ITP patients with normal level of vWF, ITP patients with decreased MA of thromboelastography

SUMMARY:
The investigators are trying to investigate the coagulation status of idiopathic (immune) thrombocytopenic purpura patients by measuring the platelet count, coagulation battery, von Willebrand factor level, thromboelastography.

DETAILED DESCRIPTION:
In patients with chronic coagulation disorder, laboratory model and clinical data have shown evidence for a rebalanced hemostasis. Previous study showed that the platelet count may not predict the risk of bleeding since the platelet count is not an indicator of platelet function. Thromboelastography may be the choice of investigation when platelet function is in question especially in patients with idiopathic (immune) thrombocytopenic purpura (ITP). Previous study have shown that maximum clot formation is the most important thromboelastography parameter in predicting bleeding in ITP patients that makes thromboelastography superior to other hemostatic tests. The investigators are trying to evaluate the rebalanced hemostasis in patients with ITP by comparing the value of platelet count, von Willebrand factor antigen level, and thromboelastography parameters.

ELIGIBILITY:
Inclusion Criteria:

* Those who visits the outpatients clinic of Samsung Medical Center with a diagnosis of idiopathic (immune) thrombocytopenic purpura (ITP)between March, 2012 and February, 2013.
* Those with age between 20 and 70 yrs old

Exclusion Criteria:

* Those with other causes of thrombocytopenia other than ITP

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who visits the outpatients clinic of Samsung Medical Center with a diagnosis of idiopathic (immune) thrombocytopenic purpura between March, 2012 and February, 2013.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
maximum clot formation | within 3 hour of blood sampling
  thromboelastography parameters performed within 3 hours of blood sampling

SECONDARY OUTCOMES:
platelet count | within 1 hours of blood sampling
  platelet count
Coagulation battery results | within 1 hour after blood sampling
  prothrombin time (%, second, INR) activated partial thromboplastin time (sec) fibrinogen level (mg/dL)
von Willebrand factor antigen | within 3 hours of blood sample
  von Willebrand factor antigen level
clotting time | within 3 hours of blood sampling
  clotting time of Thromboelastography
alpha angle | within 3 hours of blood sample
  alpha angle of thromboelastography parameter
A10, A15, A20, A25 | within 3 hours of blood sampling
  amplitude 10, 15, 20, 25 minutes (mm) of thromboelastography parameter
LY 60 | within 3 hours of blood sampling
  maximum amplitude at 60 minutes of thromboelastography parameter
CLI | within 3 hours of blood sampling
  clot lysis index of thromboelastography parameter
Maximum lysis | within 3 hours of blood sampling
  Maximum lysis of thromboelastography parameter

CONTACTS AND LOCATIONS:
Overall Officials: Gaab Soo Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea